CLINICAL TRIAL: NCT01700309
Title: Young Fit and Happy - Meaningful Physical Activity as Means to Improve Quality of Life and Prevent Weight Gain in Over-weight and Obese Adolescents. A Web-based Intervention.
Brief Title: Young, Fit and Happy. A Web-based Intervention to Prevent Obesity in Adolescents.
Acronym: YFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Sølvi Helseth, Professor, Oslo Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010/2978
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Overweight and Obesity
Keywords: Obesity prevention; Adolescent; Physical activity; Health counselling
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Treatment as usual
- Young and Active (Experimental): This arm will recieve web-based health counselling through the web-site Young and Active.
  Interventions: Behavioral: Young and Active

INTERVENTIONS:
Behavioral: Young and Active — The intervention will consist of three meetings between the adolescent, the parents and the researchers, and weekly web-based health-counselling. The adolescents will set goals and make an individual activity plan on the web-page. During the study period all activity will be registered by the adolescents. The researchers will perform weekly counseling based on Selfdetermination Theory and Motivational Interviewing. The webiste also allows for the adolescents to communicate with eacother and with the counsler through a blog.
  Arms: Young and Active

SUMMARY:
The prevalence of overweight and obesity is increasing throughout the world. Obesity is seen as one of the most important public health threats because of the significant impact of chronic conditions associated with obesity. Obesity during adolescence is a strong precursor of obesity and related morbidity in adulthood.

Interventions aimed directly at reducing weight or preventing increase in weight shows limited results on long term effects and it is shown that increase in activity has more impact on health outcome than on weight-loss. Further, weight-loss does not seem to be an appropriate measure of therapeutic interventions for growing children. The hypothesis of this study is that focusing on increasing meaningful physical activity through individual tailored counselling will have positive effects on the adolescents' fitness (health) and quality of life. Thus, the overall purpose of the study is to examine the extent to which a web-based intervention influences physical activity, fitness and quality of life in over-weight and obese adolescents Further, the aim is to explore and describe how adolescents experience being over-weight and obese, what they perceive as meaningful physical activity and finally how adolescents experience lifestyle changes as demanded in the intervention study.

DETAILED DESCRIPTION:
The target group is overweight adolescents, meaning their BMI is over or equal to the 95th percentile (BMI>25) and they should not have severe health problems as a result of their overweight. For adults, BMI (Body Mass Index; weight in kilograms divided by the square of height in meters) values at or above 25 indicate overweight and a BMI at or above 30 defines obesity. No such generally accepted definitions exist for children and adolescents. However, international standardized cut points have been proposed, among others by Cole et al (2000) and experts support the use of BMI cutoff points for children. The cut points proposed by Cole et al (2000) are widely used and take age, gender and sex into consideration in the estimation. The focus is primarily to prevent a negative development, and the aim is that the school health service in the future might implement a modified version of this strategy for working with overweight adolescents.

The design of the study is a complex intervention study with a multi-method design, consisting of a quasi-experimental trial and a qualitative study. The sample will be drawn from schools in Oslo. Overweight adolescents will be selected and placed in the intervention group or control group respectively. The sampling will be based on objective measures of weight and height and using Cole's index to define overweight and obesity. Weight and height will be measured by the school nurse and will be coordinated with her regular meetings with the adolescents in 8th grade.. The study group will receive the web-based intervention and the control group will receive standard care. At baseline, 3 months and 1 year both the experimental group and the control group will be measured at relevant variables. In the qualitative part of the study, in depth interviews with the adolescents in the intervention group will be performed and they will write daily unstructured blogs on the web. The sampling procedure for the qualitative part of the study will follow the sampling procedure of the intervention study. From the intervention group, a strategic or purposive sample of adolescents will be asked to participate in the qualitative part (Gerrish and Lacey 2006). A sample of maximum variation according to gender and sosio-demographic variables is intended. Sampling continues until saturation is reached and the adolescents will be interviewed in depth before the intervention starts, further at 3 and 12 months after the intervention is ended.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese adolescents in 8th grade
* BMI is over or equal to the 95th percentile (BMI>25 according to Cole's index)(height and weight measured by the school nurse)
* school population

Exclusion criteria

* not have severe health problems as a result of their overweight
* not be in another treatment program

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fitness | One year
  It Hypothesised that weekly individual web-counseling will motivate overweight and obese adolescents to increased physical activity. Further we assume that increased physical activity will improve the adolescents' fitness.
  Fitness is measured with a maximal multistage 20 m shuttle run test (Leger et al., 1988)

SECONDARY OUTCOMES:
Quality of Life | one year
  It is our assumption that weekly individual web-counseling, based on theories of coping and motivation, will motivate overweight and obese adolescents to increased physical activity. Further we assume that increased physical activity will improve the adolescents' fitness (health) and their quality of life.
  Measured with Kidscreen 52.

OTHER OUTCOMES:
Motivation for Physical activity and exercise, BMI, Self-efficacy | One Year
  Motivation for Physical activity and exercise measured by the Behavioural Regulation In Exercise Questionnaire (BREQ2). BMI is calculated based on objective measures of height and weight. Self-efficacy is measured with Schwarzer 8 item questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sølvi Helseth, PhD, Principal Investigator — Oslo Metropolitan University
Locations (2):
- Norway (2):
  - Oslo and Akershus University College, Oslo
  - Norwegian School of Sport Sciences, Oslo

REFERENCES:
- [Derived] Sundar TKB, Londal K, Lagerlov P, Glavin K, Helseth S. Overweight adolescents' views on physical activity - experiences of participants in an internet-based intervention: a qualitative study. BMC Public Health. 2018 Apr 4;18(1):448. doi: 10.1186/s12889-018-5324-x. PMID 29618327
- [Derived] Riiser K, Londal K, Ommundsen Y, Smastuen MC, Misvaer N, Helseth S. The outcomes of a 12-week Internet intervention aimed at improving fitness and health-related quality of life in overweight adolescents: the Young & Active controlled trial. PLoS One. 2014 Dec 5;9(12):e114732. doi: 10.1371/journal.pone.0114732. eCollection 2014. PMID 25478791